CLINICAL TRIAL: NCT05747794
Title: AIPAC-003 (Active Immunotherapy and PAClitaxel): a Randomized, Double-blind, Placebo-controlled Phase 3 Trial Testing Eftilagimod Alpha (soluble LAG-3) in HER2-neg/low Metastatic Breast Cancer Patients Receiving Paclitaxel, Following an Open-label Dose Optimization
Brief Title: Study in Metastatic Breast Cancer Patients Receiving Eftilagimod Alpha or Placebo in Combination with Paclitaxel Chemotherapy
Acronym: AIPAC-003
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Immutep S.A.S. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIPAC-003; 2022-003323-17 (EudraCT Number)
Record Dates: First submitted 2023-02-02; First posted 2023-02-28 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — soluble LAG-3 protein, human; Paclitaxel

STUDY DESIGN:
Intervention Model Description: This trial consists of an open-label dose optimization lead-in component (phase 2) followed by a double-blinded, randomized, placebo-controlled phase 3 component.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- open label lead-in (phase 2): eftilagimod alpha 30mg + paclitaxel (Experimental): eftilagimod alpha 30mg s.c. + 80mg/m^2 paclitaxel i.v. (same-day administration): The trial consists of a chemo-immunotherapy (chemo-IO) phase followed by an immunotherapy (IO)-phase. The chemo-IO phase consists of a planned 6 cycles of 4 weeks (28 days each) that may be longer or shorter depending on chemo tolerance. The IO-phase is planned to follow the chemo-IO phase. A maximum of 13 cycles (approx. 12 months) of treatment is planned.
  Interventions: Biological: eftilagimod alpha; Drug: Paclitaxel
- open label lead-in (phase 2): eftilagimod alpha 90mg + paclitaxel (Experimental): eftilagimod alpha 90mg s.c. + 80mg/m^2 paclitaxel i.v. (same-day administration): The trial consists of a chemo-immunotherapy (chemo-IO) phase followed by an immunotherapy (IO)-phase. The chemo-IO phase consists of a planned 6 cycles of 4 weeks (28 days each) that may be longer or shorter depending on chemo tolerance. The IO-phase is planned to follow the chemo-IO phase. A maximum of 13 cycles (approx. 12 months) of treatment is planned.
  Interventions: Biological: eftilagimod alpha; Drug: Paclitaxel
- Phase 3: eftilagimod alpha + paclitaxel (Experimental): eftilagimod alpha s.c. (OBD) + 80mg/m^2 paclitaxel i.v. (same-day administration): The trial consists of a chemo-immunotherapy (chemo-IO) phase followed by an immunotherapy (IO)-phase. The chemo-IO phase consists of a planned 6 cycles of 4 weeks (28 days each) that may be longer or shorter depending on chemo tolerance. The IO-phase is planned to follow the chemo-IO phase. A maximum of 13 cycles (approx. 12 months) of treatment is planned.
  Interventions: Biological: eftilagimod alpha; Drug: Paclitaxel
- Phase 3: placebo + paclitaxel (Placebo Comparator): placebo s.c. + 80mg/m^2 paclitaxel i.v. (same-day administration): The trial consists of a chemo-immunotherapy (chemo-IO) phase followed by an immunotherapy (IO)-phase. The chemo-IO phase consists of a planned 6 cycles of 4 weeks (28 days each) that may be longer or shorter depending on chemo tolerance. The IO-phase is planned to follow the chemo-IO phase. A maximum of 13 cycles (approx. 12 months) of treatment is planned.
  Interventions: Drug: Paclitaxel; Other: placebo

INTERVENTIONS:
Biological: eftilagimod alpha — APC activator, MHC II agonist
  Other Names: IMP321; efti; LAG-3Ig; eftilagimod alfa
  Arms: Phase 3: eftilagimod alpha + paclitaxel; open label lead-in (phase 2): eftilagimod alpha 30mg + paclitaxel; open label lead-in (phase 2): eftilagimod alpha 90mg + paclitaxel
Drug: Paclitaxel — paclitaxel will be given as standard of care (chemotherapy)
Other: placebo — placebo matching eftilagimod alpha
  Other Names: placebo matching eftilagimod alpha
  Arms: Phase 3: placebo + paclitaxel

SUMMARY:
The goal of this clinical trial is to compare the safety and efficacy of eftilagimod alpha (efti) in combination with paclitaxel standard of care chemotherapy in participants with metastatic breast cancer.

The main questions it aims to answer are:

* What is the optimal biological dose (OBD) of efti in combination with weekly paclitaxel chemotherapy?
* Can efti combined with weekly paclitaxel chemotherapy prolong overall survival in participants with metastatic breast cancer if compared to weekly paclitaxel chemotherapy alone?

In the first component of the trial (phase 2, lead-in) researchers will compare two groups (different dose levels of efti in combination with standard chemotherapy) to see if the treatment is safe and well tolerated and evaluate which is the optimal biological dose. In the second component of the trial (phase 3) researchers will assess if the treatment of metastatic breast cancer with the optimal biological dose of efti in combination with paclitaxel is superior compared to chemotherapy alone (placebo-controlled).

The treatment concept of each trial component consists of a chemo-immunotherapy phase followed by an immunotherapy phase. In the first phase participants will be treated with efti plus paclitaxel chemotherapy or placebo plus paclitaxel chemotherapy. After completion of the chemotherapy per standard of care, participants will be treated with the study agent alone.

DETAILED DESCRIPTION:
The AIPAC-003 trial consists of an open-label dose optimization lead-in component followed by a double-blinded, randomized, placebo-controlled phase 3 component.

The main objectives of the dose optimization lead-in (phase 2) are to evaluate and compare the safety and tolerability of 2 different dose levels of efti (30 mg and 90 mg) combined with paclitaxel, and to define the optimal biological dose (OBD) of efti in combination with weekly paclitaxel for the phase 3 part of the trial. Recruitment to the dose-optimization lead-in will be considered complete when 29 participants per cohort are randomized and considered evaluable for OBD analysis.

The main objective of the phase 3 is to demonstrate that overall survival (OS) is superior in participants treated with efti combined with weekly paclitaxel compared to weekly paclitaxel plus placebo. Approximately 771 participants will be randomized 2:1 to Arm A (active arm): paclitaxel + efti at OBD and Arm B (control arm): paclitaxel + placebo. The exact patient population will be defined after determination of the OBD.

The duration of the trial will be approximately 24 months for the dose optimization lead-in component and 60 months for the phase 3 component. The phase 3 will start prior to the completion of the phase 2 (once the OBD has been defined).

It is planned to conduct the trial at up to 20 sites in up to 4 countries across North America and Europe for the lead-in and at up to 150 sites in up to 25 countries across North America, Europe, Latin America and the Asian Pacific region for the phase 3.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic HR+ positive (estrogen receptor positive and/or progesterone receptor positive) or hormone receptor negative (HR˗), and HER2-neg breast adenocarcinoma, histologically proven by biopsy on the last available tumor tissue
* Participants with HR+ metastatic breast cancer (MBC) who progressed on or after ≥1 line of endocrine based therapy and are indicated to receive chemotherapy for metastatic disease
* Participants with HR- MBC (i.e. triple-negative breast cancer [TNBC]) who are indicated to receive paclitaxel chemotherapy without PD 1/PD-L1 therapy in the 1st line setting for metastatic disease
* ECOG performance status 0-1
* Expected survival longer than three months

Exclusion Criteria:

* Prior chemotherapy for metastatic breast adenocarcinoma
* Participants with HR+ MBC who have received <1 line of ET based therapy in the metastatic setting
* Participants with HR+ MBC who are not primary or secondary resistant to ET-based therapy and would be candidates to ET based therapy as per applicable treatment guidelines
* TNBC participants who are candidates for PD-1/PD-L1 therapy in combination with chemotherapy
* Disease-free interval of less than twelve months from the last dose of adjuvant chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 849 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Determination of Overall survival (OS) | Until trial end, death, withdrawal of consent or lost to follow-up, assessed up to 60 months
Determination of the Optimal Biological Dose (OBD) | Up to 15 months
Frequency of adverse events (AEs) | Up to 15 months
Severity of adverse events (AEs) | Up to 15 months
Duration of adverse events (AEs) | Up to 15 months
Occurrence of dose-limiting toxicities (DLTs) | Up to 15 months
Occurrence of clinically relevant abnormalities in vital signs | Up to 15 months
Occurrence of clinically relevant abnormalities in physical examinations | Up to 15 months
Occurrence of clinically relevant abnormalities in 12-lead ECGs | Up to 15 months
Occurrence of clinically relevant abnormalities in safety laboratory assessments | Up to 15 months

SECONDARY OUTCOMES:
Determination of Progression Free Survival (PFS), based on RECIST, v1.1 | Until occurrence of progressive disease, or the start of any further next line anticancer treatment, or until the end of the trial for any other reason, assessed up to 60 months
Evaluation of Objective Response Rate (ORR) based on RECIST v1.1 | Until occurrence of progressive disease, or the start of any further next line anticancer treatment, or until the end of the trial for any other reason, assessed up to 60 months
Changes from baseline in quality of life (QOL) as assessed by questionnaire of European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 | Up to 13 months
  EORTC QLQ-C30 is a 30-item self-administered cancer specific questionnaire designed to measure QOL in the cancer population
PK parameter: area under the curve (AUC) (dose optimization lead-in only) | Up to 4 months
PK parameter: peak serum concentration (Cmax) (dose optimization lead-in only) | Up to 4 months
PK parameter: time to reach Cmax (tmax) (dose optimization lead-in only) | Up to 4 months
PK parameter: systemic clearance (CL) (dose optimization lead-in only) | Up to 4 months
PK parameter: elimination half-life (t1/2) (dose optimization lead-in only) | Up to 4 months
PK parameter: volume of distribution (VD) (dose optimization lead-in only) | Up to 4 months

CONTACTS AND LOCATIONS:
Locations (22):
- United States (5):
  - The Oncology Institute, Whittier, California
  - The George Washington University Cancer Center, Washington D.C., District of Columbia
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - Oncology Consultants, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (6):
  - AZ Sint-Jan Brugge Oostende av, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hopital de Charleroi - Hopital Notre Dame, Charleroi
  - Universitair Ziekenhuizen Antwerpen, Edegem
  - Centre Hospitalier de l'Ardenne, Libramont
  - Clinique Saint-Pierre- Ottignies, Ottignies-Louvain-la-Neuve
- ARENSIA Exploratory Medicine LLC, Tbilisi, Georgia
- ARENSIA Exploratory Medicine Phase I Unit, Chisinau, Moldova
- Spain (9):
  - Institut Català d'Oncologia, Badalona
  - VHIO - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Parc Taulí Hospital Universitari, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Jaén, Jaén
  - Unidad Ensayos Clínicos Oncología Fundació IRB Lleida, Lleida
  - START Madrid - FJD, Hospital Fundación Jiménez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No